CLINICAL TRIAL: NCT06906393
Title: The Physiological Adaptations to 4-s Sprint Interval Training at Different Intensities of Maximal Power
Brief Title: Adaptations to 4-s Sprint Interval Training at Different Intensities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004970
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Fitness
Keywords: exercise; cardiovascular fitness; sprint; interval training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training group 50% Pmax (Active Comparator)
  Interventions: Behavioral: Preventive treatment
- Training group 75% Pmax (Experimental)
  Interventions: Behavioral: Preventive treatment
- Training group All-out Pmax (Experimental)
  Interventions: Behavioral: Preventive treatment

INTERVENTIONS:
Behavioral: Preventive treatment — 4-second Sprint Interval Training (SIT) over 8 weeks to improve cardiovascular health.

SUMMARY:
The purpose of this study is to investigate the chronic effects (i.e., 8 weeks, 3 times per week) of training at 50% and 75% of maximal power with 4-s sprint interval training on physiological adaptations. We previously examined the effect of training with an all-out intensity (i.e., 100% of maximal power) and reported increases in cardiorespiratory fitness. Now, we propose to examine the effects of a lower exercise intensity domains on cardiovascular fitness and its ability to stimulate the cardiorespiratory system. We hypothesize that training at 50% and 75% of maximal power will improve cardiorespiratory fitness similar to our previous findings while reducing the rate of perceived exertion during the exercise session. It is anticipated that the group engaged in training at 75% of maximal power will experience greater improvements in comparison to the group training at 50%.

DETAILED DESCRIPTION:
Background Sprint interval training (SIT) is a well-established method for improving cardiovascular and anaerobic performance. While most research focuses on all-out efforts, less is known about the effects of submaximal sprint intensities on these adaptations. This study examined how training at 50%, 75%, and all-out (85%) of maximal anaerobic power (Pmax) influences aerobic capacity and anaerobic power over an 8-week training period.

Methods

Participants: 24 recreationally active adults (12 females, 12 males) were randomly assigned to one of three training groups:

50% Pmax

75% Pmax

All-out (85% Pmax)

Training Protocol: Participants completed three sessions per week for eight weeks. Each session consisted of thirty 4-second sprints on a cycling ergometer, totaling 10 minutes per session.

Measurements: Peak oxygen consumption (VO₂peak) and maximal anaerobic power (Pmax) were assessed before and after the training program.

ELIGIBILITY:
Inclusion Criteria:

* Young (18-30),
* Healthy,
* Recreationally active, but untrained (not meeting ACSM's recommendations of 150 min/week of moderate-vigorous aerobic exercise)

Exclusion Criteria:

* Cardiovascular disease
* Smoking
* Subjects who were exercising regularly (>75 min/week) were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Maximal anaerobic power | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Department of Kinesiology and Health Education, the University of Texas at Austin, Austin, Texas, United States